CLINICAL TRIAL: NCT01804660
Title: A One Year Longitudinal Therapeutically Non-Interventional Study of MSRV-Env Burden in Normal Population as Assessed by PCR and ELISA in Blood
Brief Title: Longitudinal Therapeutically Non-interventional Study of MSRV-Env Burden in Normal Population
Acronym: CONTROL
Status: Completed | Type: Observational
Sponsor: GeNeuro Innovation SAS (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Other Study IDs: GN-E-003
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis (MS); Multiple Sclerosis associated RetroVirus (MSRV); MSRV envelop protein (MSRV-Env); Temelimab
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and PBMC.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 25 healthy volunteers: No study treatments administered
  Interventions: Other: No study treatments administered

INTERVENTIONS:
Other: No study treatments administered

SUMMARY:
This study intends to explore the levels of MSRV expression by analyzing the levels of MSRV transcripts in blood, as well as the levels of the MSRV-Env protein in serum in the normal population. This study is important for establishing a baseline to analyze results obtained in MS patients (another dedicated study is performed in parallel in MS patients). The study will be conducted over one year in a cohort of healthy subjects. The MSRV RNA level, MSRV-Env protein levels, reverse transcriptase activity, inflammatory markers assessed by cytokines levels will be analysed to define control levels in the normal population and their variation during one year. The data obtained in this study in healthy controls will be compared to those obtained in a parallel similar study, GN-E-002, conducted in different types of MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Signature of an informed consent;
* Male or female between 18 and 60 years of age.

Exclusion Criteria:

* Positive serology for hepatitis B or C or HIV;
* Acute infection at inclusion;
* Severe psychiatric disorder, neurological, inflammatory, or autoimmune disease;
* Pregnancy or breastfeeding;
* Heavy smokers i.e. more than 10 cigarettes per day;
* History of alcohol or drug abuse in the last 3 years;
* Participation in a clinical trial (within the last 3 months).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Blood donors coming for regular blood draw in the center of transfusion.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Establish a control value for the levels of MSRV expression in the normal population over time | 1 year
  Establish a control value for the levels of MSRV expression in the normal population over time using 3 approaches:
  * MSRV transcripts in PBMC;
  * MSRV transcripts in plasma;
  * MSRV-Env protein in serum.

SECONDARY OUTCOMES:
Inflammatory markers and reverse transcriptase activity in blood. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Etablissement Français du Sang Rhône Alpes - 1 route de Taninges, Annemasse, France